CLINICAL TRIAL: NCT05879523
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Effects of Food on the Pharmacokinetics of HRS-1893 Tablets After Single and Multiple Ascending Oral Doses in Healthy Volunteers and Patients With Obstructive Hypertrophic Cardiomyopathy
Brief Title: A Trial of HRS-1893 in Healthy Volunteers and Patients With Obstructive Hypertrophic Cardiomyopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-1893-101
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Intervention Model Description: HRS-1893 compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HRS-1893 for single ascending dose (SAD) cohorts (Experimental): Subjects will be assigned to one of 6 planned dose cohorts and receive single dose of HRS-1893
  Interventions: Drug: HRS-1893
- Placebo comparator for SAD cohorts (Placebo Comparator): Subjects will be assigned to one of 6 planned dose cohorts and receive single dose of placebo comparator
  Interventions: Drug: Placebo
- HRS-1893 for multiple ascending dose (MAD) cohorts (Experimental): Subjects will receive multiple doses of 2-4 planned dose cohorts and receive single dose of placebo comparator for MAD cohorts
  Interventions: Drug: HRS-1893

INTERVENTIONS:
Drug: HRS-1893 — subcutaneous, single dose, multiple doses
  Arms: HRS-1893 for multiple ascending dose (MAD) cohorts; HRS-1893 for single ascending dose (SAD) cohorts
Drug: Placebo — subcutaneous, single dose, multiple doses
  Arms: Placebo comparator for SAD cohorts

SUMMARY:
The purpose of this phase Ⅰ study is to evaluate the safety, tolerability and pharmacokinetics of HRS-1893 in healthy volunteers and patients with obstructive hypertrophic cardiomyopathy

ELIGIBILITY:
Inclusion Criteria:

1. Understand the study procedures and methods, voluntarily participate in the study, comply with study requirements, and sign the written informed consent form (ICF)
2. Male or female aged 18-55（adult healthy volunteers）or 18-85 (oHCM patients).
3. Body mass index (BMI) between 19 and 28 kg/m2.
4. Normal Electrocardiogram (ECG)

Exclusion Criteria:

1. History of persistent tachyarrhythmia and syncope;
2. A history of stomach or bowel surgery or excision (e.g. appendectomy, hernia repair, and/or cholecystectomy);
3. Positive results of hepatitis B surface antigen, hepatitis C antibody, syphilis antibody and human immunodeficiency virus antibody.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
incidence of adverse event (AE), serious adverse event (SAE) | Start of Treatment to end of study (approximately 34 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided